CLINICAL TRIAL: NCT02812225
Title: Non-blinded Data Collection Study of Concussion Using the BrainPulse(TM)
Status: Completed | Type: Observational
Sponsor: Jan Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: JMC-1502
Record Dates: First submitted 2016-06-20; First posted 2016-06-24 (Estimated); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Brain Concussion; Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- BrainPulse: BrainPulse recordings will be obtained from patients when they come in to the ED after a trauma event. BrainPulse recordings will be also obtained from those subjects who also consent for follow-up.
  Interventions: Device: BrainPulse

INTERVENTIONS:
Device: BrainPulse — Jan Medical's BrainPulse measures the brain motion caused by pulsatile blood flow from the cardiac cycle, referred to as the BrainPulse signal. The BrainPulse measures skull acceleration in response to the brain motion using an array of sensors placed on the head.
  Other Names: BrainPulse 1100

SUMMARY:
The multi-center study evaluates BrainPulse recordings from subjects with a suspected or confirmed concussion to improve a concussion detection algorithm. Subjects may also consent for a 5 additional follow-ups over a 21-day period to compare the progression of change in their BrainPulse recordings.

DETAILED DESCRIPTION:
The primary objective of this study is to collect un-blinded BrainPulse recordings from youth and adults that have a confirmed diagnosis of concussion per protocol guidelines in order to improve a concussion detection algorithm previously developed by Jan Medical, Inc. In order to gather sufficient variability, subjects with both confirmed concussion and suspected concussion will be included in the study as long as they meet eligibility criteria. BrainPulse recordings from subjects with suspected concussion will be compared to the recordings of subjects diagnosed with concussion. Subjects will be followed for 21 days after the initial injury with BrainPulse recordings to study the subject's recovery process. The symptomatic evaluation, physical examination, and BrainPulse recordings will be entered in a database to assess clinical outcome and device utilization.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 5 years old
2. Suspected or confirmed concussion by medical professional
3. Not more than 3 days since injury/trauma event
4. Willing and able to participate in all required study evaluations and allow access to medical testing and records
5. Signed informed consent/assent, and/or have a legally authorized representative willing to provide informed consent on behalf of the subject
6. Demonstrates a minimum of 3 of the following symptoms:

   * Headache
   * Pressure in head
   * Dizziness
   * Neck pain
   * Fatigue/ low energy
   * Nausea or vomiting
   * Irritability
   * Difficulty in concentrating/performing tasks
   * Memory impairment
   * Insomnia
   * Reduced tolerance to stress
   * Sensitivity to light
   * Difficulty balancing
   * Blurred vision
   * Confusion
   * More emotional than usual
   * Sadness
   * Nervous/Anxious
   * Vacant stare
   * Delayed verbal/motor response
   * 'Feeling like in a fog'
   * 'Don't feel right'

Exclusion Criteria:

1. Wound or open laceration on the head in the area of one of the BrainPulse sensors that would impede use of the BrainPulse device
2. Any serious medical condition that in the opinion of the medical professional would impair ability to provide informed consent/assent or otherwise disqualify a patient from participation
3. Currently participating in or planning to participate in another clinical study during the course of the current clinical study
4. Implantation of any medical device in head (e.g. ventriculoperitoneal shunt)

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients presenting to a hospital emergency department with a mechanism of injury and clinical presentation that is consistent with concussion
Sampling Method: Non-Probability Sample
Enrollment: 406 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Number of BrainPulse recordings from suspected and confirmed concussed subjects | Through study completion, expected to be 1 year
  The primary endpoint is to enroll and record BrainPulse signals from 500 subjects with a suspected concussion. To gather sufficiently diverse data, at least 300 participants will have had a confirmed diagnosis of concussion. The data will be used to improve the algorithm for aiding in the diagnosis of concussion.

SECONDARY OUTCOMES:
Specificity: Percentage of BrainPulse recordings from suspected concussed subjects that do not have the signal pattern seen within BrainPulse recordings from confirmed concussed subjects | Through study completion, expected to be 1 year
  The secondary endpoint is to compare the BrainPulse readings from patients with confirmed concussion with patients with a suspected concussion in order to study the differences and similarities between the signals. The specific signal patterns observed from confirmed concussed subjects' BrainPulse recordings will be evaluated against the BrainPulse recordings from suspected concussed subjects who are later confirmed to not have a concussion and the percentage of such subjects will be evaluated as part of the secondary outcome. This can be seen as a specificity evaluation.

OTHER OUTCOMES:
Average number of days the signal pattern seen within BrainPulse recordings from confirmed concussed subjects from the initial recording persist over the course of the 21 day follow up period. | Through study completion, expected to be 1 year
  The tertiary endpoint is to assess the differences in BrainPulse recordings between the initial visit and each subsequent follow-up visit to better understand the recovery process post concussion.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Beth Israel Deconess Medical Center Emergency Medicine, Boston, Massachusetts
  - University of Cincinnati, Department of Emergency Medicine, Cincinnati, Ohio
  - Mountain States Health Alliance, Johnson City, Tennessee

IPD SHARING:
Plan to Share IPD: No
All primary and secondary outcome measures will be made available within 6 months of study completion.

REFERENCES:
- [Background] Auerbach PS, Baine JG, Schott ML, Greenhaw A, Acharya MG, Smith WS. Detection of concussion using cranial accelerometry. Clin J Sport Med. 2015 Mar;25(2):126-32. doi: 10.1097/JSM.0000000000000117. PMID 25010149
- [Background] Smith WS, Browne JL, Ko NU. Cranial Accelerometry Can Detect Cerebral Vasospasm Caused by Subarachnoid Hemorrhage. Neurocrit Care. 2015 Dec;23(3):364-9. doi: 10.1007/s12028-015-0118-9. PMID 25761424
- [Derived] Coscia A, Stolz U, Barczak C, Wright N, Mittermeyer S, Shams T, Epstein S, Kreitzer N. Use of the Sports Concussion Assessment Tool 3 in Emergency Department Patients With Psychiatric Disease. J Head Trauma Rehabil. 2021 Sep-Oct 01;36(5):E302-E311. doi: 10.1097/HTR.0000000000000648. PMID 33656471